CLINICAL TRIAL: NCT02601560
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single- Ascending Doses of MEDI6012 in Subjects With Stable Coronary Artery Disease
Brief Title: To Evaluate Safety, Pharmacokinetics and Pharmacodynamics of MEDI6012 in Subjects With Stable Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D5780C00002
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; CAD
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- MEDI6012 24 mg IV (Experimental): Participants received a single IV dose of 24 mg MEDI6012 on Day 1.
  Interventions: Biological: MEDI6012
- MEDI6012 80 mg IV (Experimental): Participants received a single IV dose of 80 mg MEDI6012 on Day 1.
  Interventions: Biological: MEDI6012
- MEDI6012 240 mg IV (Experimental): Participants received a single IV dose of 240 mg MEDI6012 on Day 1.
  Interventions: Biological: MEDI6012
- MEDI6012 800 mg IV (Experimental): Participants received a single IV dose of 800 mg MEDI6012 on Day 1.
  Interventions: Biological: MEDI6012
- MEDI6012 80 mg SC (Experimental): Participants received a single SC dose of 80 mg MEDI6012 on Day 1.
  Interventions: Biological: MEDI6012
- Placebo Intravenous (IV) (Placebo Comparator): Participants received a single IV dose of placebo matched to MEDI6012 on Day 1 of the study.
  Interventions: Biological: Placebo IV
- MEDI6012 600 mg SC (Experimental): Participants received a single SC dose of 600 mg MEDI6012 on Day 1.
  Interventions: Biological: MEDI6012
- Placebo Subcutaneous (SC) (Placebo Comparator): Participants received a single SC dose of placebo matched to MEDI6012 on Day 1 of the study.
  Interventions: Biological: Placebo SC

INTERVENTIONS:
Biological: MEDI6012 — Participants received a single IV (24, 80, 240, and 800 mg) and SC (80 and 600 mg) MEDI6012 doses on Day 1.
  Arms: MEDI6012 24 mg IV; MEDI6012 240 mg IV; MEDI6012 600 mg SC; MEDI6012 80 mg IV; MEDI6012 80 mg SC; MEDI6012 800 mg IV
Biological: Placebo SC — Participants received a single SC dose of placebo matched to MEDI6012 on Day 1 of the study.
  Arms: Placebo Subcutaneous (SC)
Biological: Placebo IV — Participants received a single IV dose of placebo matched to MEDI6012 on Day 1 of the study.
  Arms: Placebo Intravenous (IV)

SUMMARY:
This is a Phase 2a randomized, double-blind (subject/investigator blinded, MedImmune unblinded), placebo-controlled, dose-escalation study to evaluate the safety, PK/PD, and immunogenicity of single IV and SC MEDI6012 doses in adult subjects with stable CAD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 40 - 75 years old
* History of Stable CAD
* Currently receiving statin as standard of care

Exclusion Criteria:

* Severe angina pectoris symptoms
* High-risk coronary or carotid artery disease that will likely require surgical or percutaneous intervention during the study period
* Hospitalization for heart failure within 12 months prior to screening
* Uncontrolled Hypertension
* Within 6 months prior to screening, a history of ACS or hospitalization for heart failure
* Clinically significant abnormalities in rhythm, conduction or morphology of ECG
* Subjects with transplanted heart, left ventricular assist device, implanted pacemaker, implantable cardioverter defibrillator, or cardiac resynchronization therapy
* Untreated life-threatening ventricular arrhythmias
* History, within 12 months prior to screening, of myocarditis or restrictive pericarditis, or hemodynamically significant valvular hear disease or aortic disease
* Undergone major surgery with in 3 months prior to screening or has planned major surgery during the study period

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2016-08-20 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Research Site, Anniston, Alabama
  - Research Site, Jacksonville, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Durham, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, San Antonio, Texas
  - Research Site, Falls Church, Virginia

REFERENCES:
- [Derived] George RT, Abuhatzira L, Stoughton SM, Karathanasis SK, She D, Jin C, Buss NAPS, Bakker-Arkema R, Ongstad EL, Koren M, Hirshberg B. MEDI6012: Recombinant Human Lecithin Cholesterol Acyltransferase, High-Density Lipoprotein, and Low-Density Lipoprotein Receptor-Mediated Reverse Cholesterol Transport. J Am Heart Assoc. 2021 Jul 6;10(13):e014572. doi: 10.1161/JAHA.119.014572. Epub 2021 Jun 14. PMID 34121413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 230 participants were screened in the study from 07-Dec-2015 to 13-Jan-2017 at 8 sites in the United States of America.
Pre-assignment Details: Out of 230 participants, 182 participants were considered screen failures. The remaining 48 participants were randomized to receive the study drug. The 1600 mg dose was omitted based on a greater than expected pharmacodynamics effects at lower doses.
Groups:
- MEDI6012 24 Milligram (mg) IV: Participants received a single IV dose of 24 mg MEDI6012 on Day 1.
Period: Overall Study
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Started | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6 | 4 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: As-treated Population: All participants who received any amount of study drug were included in this population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (6.5) | 59.8 (7.0) | 60.0 (6.4) | 63.5 (5.4) | 65.8 (8.2) | 62.0 (9.3) | 71.3 (3.4) | 66.5 (4.7) | 64.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 2 | 1 | 1 | 0 | 1 | 9
  Male | 7 | 6 | 3 | 4 | 5 | 3 | 6 | 5 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are the events between first dose of study drug and up to 57 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline (Day 1) up to Day 57
Population: As-treated Population: All participants who received any amount of study drug were included in this population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Participants
  TEAEs | 3 | 2 | 5 | 2 | 4 | 2 | 3 | 4
  TESAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With TEAEs Related to Electrocardiogram (ECG) Evaluations
Description: TEAEs observed in participants with clinically significant ECG abnormalities were assessed. TEAEs are the events between first dose of study drug and up to 57 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline (Day 1) up to Day 57
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With TEAEs Related to Vital Sign Parameters
Description: TEAEs observed in participants with clinically significant vital signs abnormalities were assessed. Vital signs parameters included blood pressure, respiration rate, pulse, pulse oximetry, and body temperature.
Time Frame: Baseline (Day 1) up to Day 57
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With TEAEs Related to Clinical Laboratory Evaluations
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Laboratory evaluations (haematology, serum chemistry and urinalysis) of blood and urine samples were performed.
Time Frame: Baseline (Day 1) up to Day 57
Population: As-treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

5. Primary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hours (Hrs) (AUC [0-96 Hrs]) for High-Density Lipoprotein-Cholesterol (HDL-C)
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of HDL-C.
Time Frame: Pre-dose, 12, 24, 48, 72 and 96 hrs post-dose Day 1 for IV and SC dose; additional within 5 minutes after completion of infusion, 4 and 8 hrs post-dose Day 1 (IV cohorts only)
Population: As-treated Population.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
milligrams per deciliter (mg/dL) | -49.1 (120.0) | 728.3 (334.2) | 1639.9 (631.7) | 3035.0 (439.1) | 5318.3 (1674.3) | -113.5 (289.4) | 422.4 (395.7) | 2844.7 (1219.1)
Statistical Analysis 1: Comparison: Placebo Intravenous (IV) vs MEDI6012 24 Milligram (mg) IV; Test type: Superiority or Other; p = 0.095, ANCOVA
Statistical Analysis 2: Comparison: Placebo Intravenous (IV) vs MEDI6012 80 mg IV; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Placebo Intravenous (IV) vs MEDI6012 240 mg IV; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Placebo Intravenous (IV) vs MEDI6012 800 mg IV; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Placebo Subcutaneous (SC) vs MEDI6012 600 mg SC; Test type: Superiority or Other; p = 0.440, ANCOVA
Statistical Analysis 6: Comparison: Placebo Subcutaneous (SC) vs MEDI6012 80 mg SC; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for Total Cholesterol
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of total cholesterol.
Time Frame: Pre-dose, 12, 24, 48, 72 and 96 hrs post-dose Day 1 for IV and SC dose; additional within 5 minutes after completion of infusion and 4 and 8 hrs post-dose Day 1 (IV cohorts only)
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | 13.8 (954.1) | -164.9 (1301.5) | 1925.7 (913.3) | 3639.2 (667.6) | 6990.3 (1764.0) | 82.3 (983.4) | 240.9 (494.2) | 3156.8 (1476.5)

7. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for Free Cholesterol
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of free cholesterol.
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | 38.4 (265.4) | -197.7 (338.2) | 38.9 (346.8) | 110.0 (133.9) | 434.6 (541.7) | 172.5 (76.6) | -61.5 (206.6) | -205.4 (324.5)

8. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for Cholesteryl Ester
Description: The AUC(0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of cholesteryl ester.
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | -24.6 (776.0) | 32.8 (992.6) | 1886.8 (722.8) | 3529.2 (628.3) | 6555.7 (1674.0) | -90.2 (965.4) | 302.4 (428.4) | 3362.3 (1340.5)

9. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for High-Density Lipoprotein Cholesteryl Ester
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of high density lipoprotein cholesteryl ester.
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | -50.3 (108.9) | 668.4 (263.3) | 1460.7 (584.0) | 2778.0 (416.7) | 4886.0 (1459.7) | -132.6 (253.1) | 392.7 (350.3) | 2672.5 (1115.7)

10. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for Non-High Density Lipoprotein Cholesterol
Description: The AUC(0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of non-high density lipoprotein cholesterol.
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | 63.0 (906.4) | -893.2 (1316.0) | 285.8 (1051.8) | 604.2 (659.1) | 1672.0 (1413.4) | 195.8 (809.9) | -181.5 (385.1) | 312.2 (642.4)

11. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for High-Density Lipoprotein Unesterified Cholesterol
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of high density lipoprotein unesterified cholesterol.
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | 1.2 (38.0) | 59.9 (78.9) | 179.2 (116.5) | 248.4 (37.6) | 417.1 (256.1) | 19.1 (46.6) | 29.7 (77.5) | 172.2 (156.6)

12. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for Non-High Density Lipoprotein Cholesteryl Ester
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of non-high density lipoprotein cholesteryl ester.
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | 25.8 (748.1) | -635.6 (984.0) | 426.1 (723.0) | 741.6 (590.5) | 1649.5 (1007.5) | 42.4 (791.6) | -90.3 (390.6) | 689.8 (634.5)

13. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for Non-High Density Lipoprotein Unesterified Cholesterol
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of non-high density lipoprotein unesterified cholesterol.
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | 37.2 (241.2) | -257.6 (351.8) | -140.3 (354.7) | -132.2 (139.9) | 27.8 (609.9) | 153.4 (72.9) | -91.2 (155.2) | -377.6 (280.7)

14. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) for Low Density Lipoprotein-Cholesterol (Direct)
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of low density lipoprotein cholesterol (direct).
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | 182.1 (600.9) | -473.0 (1096.4) | 83.2 (762.0) | 987.2 (453.8) | 1812.8 (1081.8) | -101.6 (854.2) | -61.7 (438.1) | 996.1 (803.5)

15. Secondary Outcome: Baseline-adjusted Area Under the Curve From Time 0 to 96 Hrs (AUC [0-96 Hrs]) Post Dose for Apolipoprotein B
Description: The AUC (0-96 hrs) is the area under the concentration-time curve from time 0 to 96 hrs of apolipoprotein B.
Time Frame: as for outcome 6
Population: As-treated population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL | 220.7 (524.7) | -795.5 (695.5) | -636.7 (682.6) | -649.5 (208.6) | -537.1 (706.2) | 97.4 (483.2) | -309.0 (270.5) | -219.0 (630.7)

16. Secondary Outcome: Change From Baseline in Serum Concentration of Pre Beta 1-High Density Lipoprotein at Day 29
Description: The change from baseline in serum concentration of pre beta 1-high density lipoprotein was estimated.
Time Frame: Baseline (Day 1) and Day 29
Population: As-treated population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
mg/dL
  Baseline (Day 1): number analyzed (Participants) | 8 | 6 | 6 | 4 | 6 | 1 | 5 | 3
  Baseline (Day 1) | 3.68 (2.24) | 1.75 (0.37) | 2.08 (1.19) | 2.53 (1.80) | 4.85 (4.01) | 3.90 (NA) — Standard deviation cannot be determined as only 1 participant was available. | 3.38 (1.48) | 1.67 (0.46)
  Change at Day 29: number analyzed (Participants) | 8 | 6 | 4 | 3 | 6 | 1 | 4 | 3
  Change at Day 29 | -0.20 (1.27) | -0.02 (0.84) | 0.13 (0.32) | 0.40 (0.62) | -1.12 (3.21) | -1.10 (NA) — Standard deviation cannot be determined as only 1 participant was available. | 1.33 (1.44) | 0.10 (0.60)

17. Secondary Outcome: Change From Baseline in Serum Concentration of Lecithin-Cholesterol Acyltransferase (LCAT) at Day 57
Description: The change from baseline in serum concentration of lecithin-cholesterol acyltransferase was estimated.
Time Frame: Baseline (Day 1) and Day 57
Population: Pharmacokinetic (PK) population: All participants in the as-treated population who had atleast one detectable LCAT serum concentration measurement.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6
mcg/mL
  Baseline (Day 1) | 1250.0 (0.0) | 1250.0 (0.0) | 1250.0 (0.0) | 1250.0 (0.0) | 1250.0 (0.0) | 1250.0 (0.0)
  Change at Day 57: number analyzed (Participants) | 1 | 0 | 0 | 2 | 1 | 0
  Change at Day 57 | 0.0 (NA) — Standard deviation cannot be determined as only 1 participant was available. |  |  | 0.0 (0.0) | 0.0 (NA) — Standard deviation cannot be determined as only 1 participant was available. |

18. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI6012
Description: The first occurrence of the maximum observed plasma concentration of MEDI6012 determined directly from the raw concentration time data.
Time Frame: Pre-dose and within 5 minutes; 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 and 168 hrs post-dose Day 1 for IV and SC dose, Day 15 and Day 29; additional 30 min after start of 1-hour infusion (IV cohorts only)
Population: PK population. PK data of MEDI6012 80 mg SC dose group was not interpretable as concentration levels were predominantly beneath the limit of quantitation (<2.5 mcg/mL).
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | MEDI6012 600 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
micrograms/milliliter (mcg/mL) | 5.02 (2.25) | 20.2 (4.15) | 73.5 (9.40) | 229 (55.4) | 22.8 (9.75)

19. Secondary Outcome: Time to Reach Concentration Maximum (Tmax) of MEDI6012
Description: The time at which Cmax of MEDI6012 was observed determined directly from raw concentration time data.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Median (Full Range); unit: hrs
Arm/Group | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | MEDI6012 600 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hrs | 1.00 (2.25) [1.00 to 1.00] | 1.00 (4.15) [1.00 to 1.50] | 1.00 (9.40) [1.00 to 2.00] | 1.00 (55.4) [1.00 to 1.50] | 48.0 (9.75) [48.0 to 72.0]

20. Secondary Outcome: Area Under the Concentration Time Curve From 0 to 168 Hrs (AUC [0-168]) of MEDI6012
Description: The area under the concentration-time curve from 0 to 168 hrs of MEDI6012.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | MEDI6012 600 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
mcg*hr/mL | 137 (55.0) | 805 (265) | 2760 (249) | 8470 (2000) | 2460 (824)

21. Secondary Outcome: Area Under the Concentration Time Curve From Time Zero to Last Quantifiable Concentration (AUC [0-last]) of MEDI6012
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUC [0-last]) of MEDI6012.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | MEDI6012 600 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
mcg*hr/mL | 46.8 (42.7) [1.00 to 1.00] | 683 (267) [1.00 to 1.50] | 2760 (249) [1.00 to 2.00] | 9020 (2760) [1.00 to 1.50] | 2460 (824) [48.0 to 72.0]

22. Secondary Outcome: Area Under the Concentration Time Curve to Infinite Time (AUC [0-inf]) of MEDI6012
Description: The area under the concentration-time curve to infinite time of MEDI6012.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | MEDI6012 600 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
mcg*hr/mL | 137 (56.1) | 887 (308) | 3030 (298) | 9510 (2720) | 3560 (732)

23. Secondary Outcome: Elimination Half Life (t1/2) of MEDI6012
Description: The t1/2 is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | MEDI6012 600 mg SC
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hrs | 17.6 (5.47) | 46.9 (17.6) | 45.7 (3.67) | 55.4 (14.2) | 89.5 (46.7)

24. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies for MEDI6012
Description: Participants were tested for immunogenicity to MEDI6012. The neutralization assay measures the capacity of participant's plasma (antibodies) to inhibit the binding of MEDI6012 to its target.
Time Frame: Day 1 (pre-dose), 15, 29 and 57
Population: Immunogenicity population: All participants in the as-treated population with at least one serum sample available for immunogenicity testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Participants
  Day 1 (predose) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Day 29: number analyzed (Participants) | 8 | 6 | 5 | 6 | 6 | 3 | 6 | 5
  Day 29 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Day 57: number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
  Day 57 |  | 0 |  |  | 2 |  | 1 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline (Day 1) throughout the treatment period and including the follow-up period (up to Day 57).
Arm/Group | Placebo Intravenous (IV) | MEDI6012 24 Milligram (mg) IV | MEDI6012 80 mg IV | MEDI6012 240 mg IV | MEDI6012 800 mg IV | Placebo Subcutaneous (SC) | MEDI6012 80 mg SC | MEDI6012 600 mg SC
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/8 | 2/6 | 5/6 | 2/6 | 4/6 | 2/4 | 3/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Intravenous (IV) (N=8) | MEDI6012 24 Milligram (mg) IV (N=6) | MEDI6012 80 mg IV (N=6) | MEDI6012 240 mg IV (N=6) | MEDI6012 800 mg IV (N=6) | Placebo Subcutaneous (SC) (N=4) | MEDI6012 80 mg SC (N=6) | MEDI6012 600 mg SC (N=6)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Medical device site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
High density lipoprotein decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Slow speech (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.